CLINICAL TRIAL: NCT03744871
Title: ASPIRE: Air Pollution: Strategies for Personalized Intervention to Reduce Exposure
Brief Title: Air Pollution: Strategies for Personalized Intervention to Reduce Exposure
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: University of Michigan (Other); Peking University (Other)
Responsible Party: Principal Investigator, Sanjay Rajagopalan, Division Chief, Cardiovascular Medicine, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 03-18-20; R01ES019616 (NIH)
Record Dates: First submitted 2018-04-27; First posted 2018-11-16 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Air Pollution
MeSH Terms: interventions — N95 Respirators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Respirator (Active Comparator): Open label use of N95 respirators (worn outdoors) (active limb, n=100)
  Interventions: Other: N95 Respirator
- No intervention (No Intervention): No respirators will be worn by the control group (control limb, n=100)

INTERVENTIONS:
Other: N95 Respirator — SiTi N95 respirator with microventilator (change twice weekly and earlier as needed).
  Arms: Respirator

SUMMARY:
Fine particulate matter < 2.5 microns (PM2.5) air pollution is a leading global risk factor for cardiovascular morbidity and mortality. PM2.5 presents a serious ongoing public health threat to patients living in highly-polluted countries (ex: China, India) where air quality is projected to remain extremely poor (far exceeding World Health Organization Air Quality Guidelines) for the foreseeable future. This study reviews the benefits of personal level intervention (wearing N95 respirator) over long term, to prevent clinical events among patients with cardiovascular disease.

DETAILED DESCRIPTION:
CLEANAIR-ACS will be an investigation within ASPIRE, that will test the ability of personal-level intervention (N95 respirators) to improve validated surrogate markers of cardio-metabolic health in patients with a recent Acute Coronary Syndrome (ACS). Patients with ACS are a vulnerable patient population with vulnerability and at risk for future cardiovascular events. This vanguard phase study in Beijing involving patients exposed to high levels of air pollution who have recently sustained an ACS event, is necessary to obtain feasibility data and gather a battery of information allowing for the appropriate design of a larger clinical outcome trial. What is more, positive results would provide critically-important information demonstrating for the first time that it is feasible to "prescribe" the use of these personal protection devices to cardiac patients, and that their usage is capable of translating into demonstrable health benefits (i.e., improved BP and insulin sensitivity) over the long-term.

The study hypothesis is that long-term personal-level interventions to reduce exposure to PM2.5 can be feasibly performed for 1-year post-acute coronary syndrome (ACS) and will result in significant improvements in validated surrogate cardiometabolic endpoints predictive of morbidity/mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >18, able to provide informed consent and willingness to complete the study protocol and measurement procedures, AND
2. Non-smoker of any type (cigarette, cigar, marijuana) during past six months (100% abstinence per self-report) and living in a non-smoking household (no person living in the household smoking at home) with confirmation of non-smoking status by urinary cotinine levels.

AND 3. A diagnosis of myocardial infarction or unstable angina 7-90 days prior to signed informed consent

Exclusion Criteria:

1. Inability for mental or physical reasons to understand and comply with the informed consent process and/or the study protocol procedures including wearing face mask (i.e: advanced COPD/lung disease requiring use of frequent inhalational or nebulizer treatments) per investigator discretion.
2. Obesity with arm circumference >18 inches preventing accurate BP determination during ABPM monitoring
3. Significant hemodynamically unstable CV disorder including uncompensated heart failure, refractory angina, uncontrolled arrhythmias, critical valvular heart disease and severe hypertension. (as further described in Appendix B) at screening
4. ESRD on dialysis or patients that have received dialysis within 14 days prior to screening
5. Subject has a history of infection with human immunodeficiency virus
6. Subject has a history of alcohol or substance abuse within the 6 months prior to the screening
7. Advanced COPD on home oxygen
8. Past diagnosis of sleep apnea either untreated or treated with CPAP
9. History of malignancy including leukemia and lymphoma (but not basal cell skin cancer, cured squamous cell cancer and localized Prostate cancer) AND/OR any severe, life-threatening disease AND/OR history of drug abuse within the last 2 years
10. Regular use of any over-the-counter drug, recreational medication including stimulants (amphetamines) and/or complimentary or herbal therapy that might impact study outcomes including BP and insulin sensitivity per investigator discretion.
11. In women of childbearing age: pregnancy, non-use of approved method of birth control, intent to get pregnant during the study period
12. Patients with passive home cigarette smoking
13. Other medical or psychosocial conditions or life circumstances that may put the subject at increased risk of participation or jeopardizes the scientific integrity of the study, as determined by the investigators

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 12 months
  Use Omron 907xl for clinic BP Measures, with 3 repeated measurements after 5 minutes after clinicians leave room (patient unattended). Averages of the 3 BP Recordings will be obtained

SECONDARY OUTCOMES:
PWV and pulse wave analysis | 12 months
  To be measured at clinic visits, with Omron used in JI Study
BP/HRV Monitoring | 12 months
  24 hour ambulatory HRV/BP will be placed when clinic BP is complete as the first clinic measure. The monitoring systems have been used in JI study previously

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States
- Peking University, Beijing, China